CLINICAL TRIAL: NCT02135016
Title: The Effect of Thoracic Epidural Anesthesia With Different Block Level on Propofol Concentration During General Anesthesia Induction
Brief Title: The Effect of Thoracic Epidural Anesthesia With Different Block Level on Propofol Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Jun Wang, professor, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20140415
Record Dates: First submitted 2014-04-30; First posted 2014-05-09 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Target Controlled Infusion (TCI); Thoracic Epidural Anesthesia; Block Level; Gastrointestinal Surgery
Keywords: effect-site concentration; propofol; thoracic epidural anesthesia
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1% lidocaine (Experimental): epidural anesthesia with 1% lidocaine 10ml before propofol TCI
  Interventions: Drug: 1% lidocaine
- 2% lidocaine (Experimental): epidural anesthesia with 2% lidocaine 5ml before propofol TCI
  Interventions: Drug: 2% lidocaine
- 0.9% normal saline (Placebo Comparator): epidural anesthesia with 0.9% normal saline 5ml before propofol TCI
  Interventions: Drug: 0.9% normal saline

INTERVENTIONS:
Drug: 1% lidocaine — epidural anesthesia with 1% lidocaine 10ml before propofol TCI
  Other Names: A
  Arms: 1% lidocaine
Drug: 2% lidocaine — epidural anesthesia with 2% lidocaine 5ml before propofol TCI
  Other Names: B
  Arms: 2% lidocaine
Drug: 0.9% normal saline — epidural anesthesia with 0.9% normal saline 5ml before propofol TCI
  Other Names: C
  Arms: 0.9% normal saline

SUMMARY:
It is a prospective, randomized, placebo-controlled study to investigate the effect of TEA with different block level on propofol concentration during general anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-II physical status,
* aged 40-60 yr,
* BMI 19-25 kg/m2,
* undergoing elective gastrointestinal surgery

Exclusion Criteria:

* patients with cardiovascular or neurological disease, drug or alcohol abuse and absolute contraindications for neuraxial blockade.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, professor, Study Director — Dept. of Anesthesiology, First Affiliated Hospital of China Medical University
Locations (1):
- Jun Wang, Shenyang, Liaoning, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1% Lidocaine | 2% Lidocaine | 0.9% Normal Saline
Started | 15 | 15 | 15
Completed | 15 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% Lidocaine | 2% Lidocaine | 0.9% Normal Saline | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (6) | 57 (7.0) | 56 (4) | 56 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 7 | 20
  Male | 8 | 9 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: The Effect-site Concentration of Propofol
Description: The effect-site concentration of propofol when loss of consciousness during propofol target-controlled infusing(TCI) induction of anesthesia.
Time Frame: The participants will be followed for the duration of anesthesia induction, an expected average of half an hour
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | 1% Lidocaine | 2% Lidocaine | 0.9% Normal Saline
Number analyzed (Participants) | 15 | 15 | 15
µg/ml | 1.51 (0.44) | 1.99 (0.37) | 2.68 (0.68)

2. Secondary Outcome: The Bispectral Index
Description: The bispectral index (BIS) of each patient will be recorded at four different time points,as follows, baseline(the awake phase before epidural anesthesia),10 mins after epidural anesthesia, 20 mins after epidural anesthesia, loss of consciousness(when the participants are lost eyelash reflex during propofol TCI induction of anesthesia). BIS values varies from 0 to 100(0, no cerebral activity; 40 to 60, general anesthesia; 60 to 85, sedated; 85 to 100, awake).
Time Frame: The participants will be followed for the duration of anesthesia induction, an expected average of half an hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Lidocaine | 2% Lidocaine | 0.9% Normal Saline
Number analyzed (Participants) | 15 | 15 | 15
units on a scale
  Baseline | 95.4 (1.4) | 95.4 (1.4) | 95.7 (1.3)
  10mins after epidural aneasthesia | 85.3 (0.7) | 85.1 (1.3) | 94.5 (0.9)
  20mins after epidural aneasthesia | 84.6 (0.9) | 83.8 (0.8) | 94.9 (1.8)
  Loss of consciousness | 65.7 (0.8) | 65.3 (2.5) | 66.1 (2.6)

3. Secondary Outcome: The Mean Blood Pressure
Description: The mean arterial pressure of each patient will be recorded at four different time points, as follows, baseline(the awake phase before epidural anesthesia), 10 mins after epidural anesthesia, 20 mins after epidural anesthesia, loss of consciousness(when the participants are lost eyelash reflex during propofol TCI induction of anesthesia).
Time Frame: The participants will be followed for the duration of anesthesia induction, an expected average of half an hour
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 1% Lidocaine | 2% Lidocaine | 0.9% Normal Saline
Number analyzed (Participants) | 15 | 15 | 15
mmHg
  Baseline | 95.4 (2.5) | 95.1 (2.1) | 95.9 (2.3)
  10mins after epidural aneasthesia | 85.9 (3.6) | 83.7 (2.6) | 95.5 (2.7)
  20mins after epidural aneasthesia | 79.3 (2.5) | 80.5 (3.0) | 96.1 (2.2)
  Loss of consciousness | 74.0 (1.4) | 74.5 (1.0) | 82.7 (1.3)

4. Secondary Outcome: The Heart Rate
Description: The heart rate of each patient will be recorded at three different four points, as follows, baseline(the awake phase before epidural anesthesia), 10mins after epidural anesthesia, 20 mins after epidural anesthesia, loss of consciousness(when the participants are lost eyelash reflex during propofol TCI induction of anesthesia).
Time Frame: The participants will be followed for the duration of anesthesia induction, an expected average of half an hour
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | 1% Lidocaine | 2% Lidocaine | 0.9% Normal Saline
Number analyzed (Participants) | 15 | 15 | 15
beats per minute
  Baseline | 71.4 (4.7) | 72.8 (3.3) | 71.3 (3.5)
  10mins after epidural aneasthesia | 69.8 (4.4) | 69.2 (3.7) | 71.3 (3.5)
  20mins after epidural aneasthesia | 68.5 (3.4) | 67.2 (3.4) | 70.3 (3.3)
  Loss of consciousness | 63.2 (1.8) | 62.3 (1.9) | 63.2 (1.8)

5. Secondary Outcome: The Block Level of Epidural Anesthesia
Description: The block level 20mins after epidural anesthesia and it is verified by the loss of sensation to alcohol swab before target controlled infusion of propofol.It is the number of block segments.The block level varies from 0 to 10(0, no block level; 1 to 5, narrow block level;6 to 10, wide block level).
Time Frame: 20 mins after epidural anesthesia
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Lidocaine | 2% Lidocaine | 0.9% Normal Saline
Number analyzed (Participants) | 15 | 15 | 15
units on a scale | 6.5 (1.0) | 4.2 (0.9) | 0 (0)

ADVERSE EVENTS:
Groups:
- Group A: epidural anesthesia with 1% lidocaine 10ml before propofol TCI
- Group B: epidural anesthesia with 2% lidocaine 5ml before propofol TCI
- Group C: epidural anesthesia with 0.9% normal saline 5ml before propofol TCI
Arm/Group | Group A | Group B | Group C
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes